CLINICAL TRIAL: NCT07260487
Title: Assessment of Anthropometric and Biochemical Indices in Predicting Metabolic Syndrome Across Obesity Classes
Brief Title: New Biomarkers for Predicting Systemic Complications in Obesity
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Elif Azize Özşahin Delibaş, Assistant Professor, Tokat Gaziosmanpasa University
Other Study IDs: 24-KAEK-008
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Metabolic Syndrome; Obesity
Keywords: metabolic syndrome; obesity; anthropometric indices; biochemical indices; cardiometabolic risk
MeSH Terms: conditions — Metabolic Syndrome; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational cross-sectional study classified participants into obesity classes (Class I: BMI 30.0-34.9, Class II: 35.0-39.9, Class III: ≥40.0 kg/m²) based on WHO criteria. Anthropometric and biochemical measurements were used to calculate a wide range of obesity-related and cardiometabolic risk indices. The aim was to analyze whether these indices could effectively predict the presence of Metabolic Syndrome (MetS), as defined by the NCEP-ATP III criteria.

DETAILED DESCRIPTION:
In this study, a comprehensive set of anthropometric, biochemical, and derived indices was utilized to assess the relationship between obesity and Metabolic Syndrome (MetS) beyond the scope of traditional measures. While Body Mass Index (BMI) served as the primary criterion for general obesity classification, it was complemented by additional indices that are considered more reflective of fat distribution and visceral adiposity. These included the Visceral Adiposity Index (VAI), Waist-to-Height Ratio (WHtR), Waist-to-Hip Ratio (WHpR), Body Adiposity Index (BAI), and Conicity Index (COI), all of which provide greater specificity in evaluating central obesity-a key factor in cardiometabolic risk.

To capture the metabolic dimension of obesity, biochemical indices such as the Triglyceride-Glucose (TyG) index were calculated, as this marker has been shown to correlate strongly with early insulin resistance and glucose homeostasis disruption. Additionally, the Lipid Accumulation Product (LAP), which combines waist circumference and triglyceride levels, was employed to estimate the extent of visceral fat accumulation and its associated metabolic burden.

To further investigate cardiovascular and atherogenic risk, several lipid-based indices were assessed, including the Atherogenic Coefficient (AC), Atherogenic Plasma Index (API), the Triglyceride-to-HDL cholesterol (TG/HDL) ratio, non-HDL cholesterol, and the Cholindex. The inclusion of these diverse indices allowed for a more nuanced and multidimensional evaluation of the associations between obesity phenotypes and MetS status, with the aim of identifying reliable predictors beyond conventional clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with obesity
* Being between the ages of 18 and 65

Exclusion Criteria:

* Having any other chronic disease (cardiovascular disease, polycystic ovary syndrome, thyroid dysfunction, asthma, etc.)
* Receiving hormone therapy
* Taking lipid-lowering medication
* Being pregnant/breastfeeding
* Having an acute infection
* Having a malignant or inflammatory disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obese adult individuals (BMI ≥30 kg/m²) aged 18-65 years who presented voluntarily to an internal medicine outpatient clinic were included in the study. Participants had no known chronic diseases, were not pregnant or breastfeeding, and were not receiving hormone therapy or lipid-lowering treatment. Individuals with cardiovascular disease, thyroid dysfunction, polycystic ovary syndrome, malignancy, inflammatory disease, acute infection, or other metabolic disorders were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) was used to classify levels of obesity. | Directly taken by trained staff during face-to-face assessments.
  BMI is an anthropometric parameter obtained by dividing body weight in kilograms by the square of height in metres (kg/m²). According to the World Health Organization (WHO) classification, individuals with a BMI of less than 18.5 kg/m² are underweight; those with a BMI between 18.5 and 24.9 kg/m² are of normal weight; those with a BMI between 25.0 and 29.9 kg/m² are overweight (pre-obese); and those with a BMI between 30.0 and 34.9 kg/m² are classified as class 1 obese (moderate); those between 35.0-39.9 kg/m² are class 2 obese (severe); and those ≥40.0 kg/m² are class 3 obese (morbid)
MetS was diagnosed according to National Cholesterol Education Program - Adult Treatment Panel III (NCEP-ATP III) criteria. | Anthropometric measurements were directly taken by trained staff during face-to-face assessments. Biochemical data were retrospectively obtained from hospital medical records.
  Five clinical parameters were evaluated accordingly: WC, FBG, HDLc, TG level and blood pressure. The following were accepted as components of MetS: WC≥102 cm in men and ≥88 cm in women; TG level ≥150 mg/dL; HDLc level <40 mg/dL in men and <50 mg/dL in women; blood pressure ≥130/85 mmHg; and FBG level ≥100 mg/dL. Individuals were classified as MetS (+) if at least three of the five specified parameters met the diagnostic criteria and as MetS (-) if they did not.
Waist-to-Height Ratio | Directly taken by trained staff during face-to-face assessments.
  Waist Circumference (cm) / Height (cm)
Waist-to-Hip Ratio | Directly taken by trained staff during face-to-face assessments.
  Waist Circumference (cm) / Hip Circumference (cm)
Lipid Accumulation Product | Anthropometric measurements were directly taken by trained staff during face-to-face assessments. Biochemical data were retrospectively obtained from hospital medical records.
  For men: [WC (cm) - 65] × TG (mmol/L) For women: [WC (cm) - 58] × TG (mmol/L)
Visceral Adiposity Index | Anthropometric measurements were directly taken by trained staff during face-to-face assessments. Biochemical data were retrospectively obtained from hospital medical records.
  For men: [WC (cm) / (39.68 + (1.88 × BMI))] × (TG / 1.03) × (1.31 / HDLc) For women: [WC (cm) / (36.58 + (1.89 × BMI))] × (TG / 0.81) × (1.52 / HDLc)
Conicity Index | Directly taken by trained staff during face-to-face assessments.
  WC (m) / [0.109 × √(Weight (kg) / Height (m))]
Body Adiposity Index | Directly taken by trained staff during face-to-face assessments.
  (Hip Circumference (cm) / [Height (m)]¹·⁵) - 18
Atherogenic Coefficient | Biochemical data were retrospectively obtained from hospital medical records.
  (Total Cholesterol - HDLc) / HDLc
Atherogenic Index of Plasma | Biochemical data were retrospectively obtained from hospital medical records.
  log10 (TG / HDLc)
TG/HDLc multiplied by Waist-to-Height Ratio combine index | Anthropometric measurements were directly taken by trained staff during face-to-face assessments. Biochemical data were retrospectively obtained from hospital medical records.
  (TG / HDLc) × WhtR
Triglyceride-Glucose Index | Biochemical data were retrospectively obtained from hospital medical records.
  ln [TG (mg/dL) × Fasting Glucose (mg/dL) / 2]

CONTACTS AND LOCATIONS:
Overall Officials: Elif A Özşahin Delibaş, Asst. Prof., Principal Investigator — Tokat Gaziosmanpaşa University, Faculty of Health Sciences, Department of Nutrition and Dietetics; Emre Y Kuyucu, Lecturer, Study Chair — Tokat Gaziosmanpaşa Üniversity, Faculty of Medicine, Department of Biostatistics
Locations (1):
- Tokat Gaziosmanpaşa University Health Research and Application Hospital, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No